CLINICAL TRIAL: NCT05175937
Title: REal World Assessment for Patients Implanted With Implantable CardioverTer DefibrIllatOr Using Bluetooth Technology
Acronym: REACTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Rapacciuolo, Principal Investigator, Federico II University
Other Study IDs: 137/21
Record Dates: First submitted 2021-11-18; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Arrhythmias; Sudden Cardiac Death; Heart Failure
Keywords: Connectivity; Remote monitoring; Cardiac Implantable Electronic Device
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APP group: Patient wearing ICD with Bluetooth® technology and smartphone APP based remote monitoring
  Interventions: Device: smartphone APP based remote monitoring
- Bedside transmitter group: Patient wearing ICD monitored remotely through a bedside transmitter
  Interventions: Device: bedside transmitter based remote monitoring

INTERVENTIONS:
Device: smartphone APP based remote monitoring — smartphone APP to monitor remotely patients implanted with ICD
  Groups: APP group
Device: bedside transmitter based remote monitoring — bedside transmitter to monitor remotely patients implanted with ICD
  Groups: Bedside transmitter group

SUMMARY:
The objective of this observational study is to assess clinical benefits of innovative features (e.g. Bluetooth technology and smartphone patient applications) in a patient population that is implanted with standard indication for implantable cardiac defibrillator.

DETAILED DESCRIPTION:
REACTION is an observational study in which patients will be followed as for clinical practice and no specific study tests/procedures will be perfprmed. After implanting a device, the patient will be assigned to an arm or to the other based on the technology of the device (bluetooth or RF) he/she wears, if he/she gives the consent to partecipate. It is not a randomized study. Patients will be enrolled consecutively until reaching the sample defined for both the arms.

ELIGIBILITY:
Inclusion Criteria:

* All patients implanted with an ICD as for standard indications
* Over 18 years of age
* Ability to provide informed consent for registry participation and be willing and able to comply with the protocol described evaluations

Exclusion Criteria:

* Subject who is, or is expected to be inaccessible for follow-up
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size will be about 1104 patients; 736 patients implanted with Bluetooth technology devices and 368 patients followed with traditional remote control.
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Adherence | 12 months
  The adherence will be measured through the following endpoints:
  • Compliance with RM quantified as percentage of patients who registered with the smartphone App
Effectiveness | 12 months
  The effectiveness based on the comparison between the App monitoring and the traditional remote control will be assessed through the following endpoints:
  • Percentage of time (days) with an active connection between device and the transmitter/smartphone app

SECONDARY OUTCOMES:
Clinical benefits in CRT area: | 12 Months
  Association between patient symptom-triggered transmissions and HF events or other clinical events detected by device diagnostics
Clinical benefits in ICD therapies | 12 months
  Clinical action taken as a result of appropriate or inappropriate ICD therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Prof Antonio Rapacciuolo,MD, PhD, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided